CLINICAL TRIAL: NCT05183503
Title: Determination of Chronic Pain, Anxiety, Depression and Perceived Stress in Adults With Temporomandibular Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Principal Investigator, Wroclaw Medical University
Other Study IDs: WMU3/2021
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Disorder; Depression; Anxiety; Pain; Stress
MeSH Terms: conditions — Temporomandibular Joint Disorders; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMD group: Patients diagnosed with TMD
  Interventions: Diagnostic Test: DC/TMD examination

INTERVENTIONS:
Diagnostic Test: DC/TMD examination — Clinical examination by examiners- experienced dentists (minimum 5 years of practice) and trained and calibrated in accordance with the protocol available on the official website of the International Network for Orofacial Pain and Related Disorders Methodology

SUMMARY:
The aim of the study was to asses levels and relationship of chronic pain, anxiety, depression and perceived stress in TMD patients .

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) is an umbrella term describing a heterogenic group of conditions concerning masticatory muscles, temporomandibular joints and surrounding hard and soft structures. Most common signs and symptoms of TMD are: orofacial pain, joint sounds such as clicking or crepitus and limitation in jaw movements . Temporomandibular disorder (TMD) is the most common cause of orofacial pain and after chronic low back pain, it is the second cause of pain and disability in the musculoskeletal system. TMDs are considered as a global problem decreasing quality of life and potentially causing chronic pain, in daily activity limitation, anxiety, depression, general health problems, decreased work productivity and can lead to work absences.

The etiology of TMD is complex, multifactorial, and in many cases unclear. The biopsychosocial model tends to cover a broad spectrum of different conditions and aspects that may play a role in TMD occurrence. It integrates biological factors (structural disorders and disturbance in function) with psychosocial aspects (emotions, cognition, behaviors, reaction to stress and pain in context of family, workplace and community) .

The prevalence of TMD is estimated between 5-12% of the general population . About 26-30% of young adults present at least one symptom of TMD . The prevalence of TMD in adults over 45 years old is estimated between 2-7%.and in patients over 65 years old 3-5% . It is often suggested that women are more often affected by TMD than men.

Many studies conducted so far indicate the existence of a strong relationship between TMD and psychosocial impairment including depression, somatization and anxiety. Patients with chronic pain condition have been found to exhibit high level of psychosocial impairments compared with painless controls . Many authors also indicate that the psychosocial factors reduce the response to the conservative treatment used among patients with TMD (occlusal splint therapy) and may increase the risk of the chronic form of this disorders.Therefore, the diagnosis of various types of psychosocial disorders among TMD patients is very important, because it will influence the appropriate clinical decisions and correct management protocol.

The available data on the relationship between TMD and psychosocial impairment contribute a lot to both the diagnosis and management of TMD. Unfortunately, the above data do not concern the prevalence and epidemiology of chronic pain, depression, anxiety and perceived stress in the polish population. Therefore, the data collected by the cited authors cannot be compared and the conclusions drawn from them cannot be used to the Polish population.

Based on these premises, the objectives of this study are to determine the level and prevalence of chronic pain, anxiety, depression and perceived stress among adult TMD patients from western Poland, and to use these data to identify and management of TMD.

A total of 219 adult patients from outpatient clinic for temporomandibular disorders participated in this retrospective study. All patients filled GCPS, GAD-7, PHQ-9 and PSS-10 questionnaires, and had TMD diagnosis based on DC/TMD examination carried out by an experienced dentist. After that statistical analysis was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study were age equal or above 18 years old and diagnosis of TMD based on DC/TMD examination form.

Exclusion Criteria:

* The exclusion were severe neurological or mental diseases, taking medications that significantly affect the neuromuscular function, alcohol and/or drug addiction, active cancer diagnosis, pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Outpatient Clinic for Temporomandibular Disorders at the Medical University in Wroclaw diagnosed with TMD using Diagnostic Criteria for Temporomandibular Disorders (DC / TMD).
Sampling Method: Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between TMD and pain assessed by Graded Chronic Pain Scale. | 1.12.2018-1.12.2021
  Each participant will fill in Graded Chronic Pain Scale. Scoring Criteria for Grading Chronic Pain Severity:
  Characteristic Pain Intensity is a 0 to 100 score derived from Questions 1 through 3:Mean (Pain Right Now, Worst Pain, Average Pain) X 10. Disability Score is 0 to 100score derived from Questions 4 through 6:Mean (Daily Activities, Social Activities, Work Activities) X 10. Disability Points: Add the indicated points for Disability Days (Question 7)and for Disability Score. Classification: GRADE 0- No TMD pain in prior 6 months. GRADE I-Low Intensity Characteristic Pain Intensity<50, Low Disability<3 Disability Point. GRADE II -High Intensity Characteristic Pain Intensity >50, LowDisability<3 Disability Points. GRADE III- High Disability3 to 4 Disability Points, Moderately Limiting (Regardless of Characteristic Pain Intensity). GRADE IV- High Disability 5 to 6 Disability Points, Severely Limiting (Regardless of Characteristic Pain Intensity).
Relationship between TMD and depression assessed by Patient Health Questionnaire - 9. | 1.12.2018-1.12.2021
  Each participant will fill in Patient Health Questionnaire - 9. PHQ-9 total score for the nine items ranges from 0 to 27.Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Relationship between TMD and perceived stress assessed by Perceived Stress Scale - 10. | 1.12.2018-1.12.2021
  Each participant will fill in Perceived Stress Scale -10. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
Relationship between TMD and anxiety assessed by Generalized Anxiety Disorder -7 | 1.12.2018-1.12.2021
  Each participant will fill in Generalized Anxiety Disorder -7 that consists of 7 items. Total score ranges 0-21 points.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical Uniwesity, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wieckiewicz M, Jenca A Jr, Seweryn P, Orzeszek S, Petrasova A, Grychowska N, Winocur-Arias O, Emodi-Perlman A, Kujawa K. Determination of pain intensity, pain-related disability, anxiety, depression, and perceived stress in Polish adults with temporomandibular disorders: A prospective cohort study. Front Integr Neurosci. 2022 Nov 2;16:1026781. doi: 10.3389/fnint.2022.1026781. eCollection 2022. PMID 36407294